CLINICAL TRIAL: NCT07027410
Title: Effect of Intermittent Normobaric Hypoxia on Executive Functions Assessed With Different Cognitive Tests in Healthy Young Subjects
Brief Title: Effect of Intermittent Normobaric Hypoxia on Executive Functions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Raquel Vaquero-Cristóbal, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 4145/2022
Record Dates: First submitted 2025-05-24; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Executive Function (Cognition); Normobaric Hypoxia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent Hypoxia Group (Experimental): Participants are exposed to a single session of intermittent normobaric hypoxia at 12% oxygen concentration (equivalent to 4400 m altitude) using the iAltitude simulator. Cognitive tests are performed before and after the hypoxia session.
  Interventions: Device: Intermittent normobaric hypoxia
- No Hypoxia Group (Other): Participants undergo the same cognitive tests without exposure to hypoxia, serving as the control condition.
  Interventions: Other: Normoxia

INTERVENTIONS:
Device: Intermittent normobaric hypoxia — Participants in the experimental group undergo a single session of intermittent normobaric hypoxia simulated by the iAltitude device. The session consists of breathing air with 12% oxygen concentration (equivalent to 4400 meters altitude) for a specified duration. Cognitive tests are administered before and after the hypoxia exposure to assess executive functions.
  Arms: Intermittent Hypoxia Group
Other: Normoxia — Participants undergo the same cognitive tests without exposure to hypoxia, serving as the control condition.
  Arms: No Hypoxia Group

SUMMARY:
The main objective of this study was to analyze the effects of an intermittent normobaric hypoxia session on executive functions assessed with different cognitive tests given to healthy young subjects. Twenty-seven healthy volunteers were divided into an experimental group (EG; n=13) and a control group (CG; n=14). The EG performed the 'Odd One Out', 'Double Trouble' and 'Monkey Ladder' tests before and after the hypoxia tolerance session (12%, 4400 m) with the iAltitude simulator. The CG completed the same tests without hypoxia exposure.

DETAILED DESCRIPTION:
The main objective of this study will be to analyze the effects of an intermittent normobaric hypoxia session on executive functions, assessed using different cognitive tests administered to healthy young subjects. A total of 27 healthy volunteers will be divided into two groups: an experimental group (EG; n=13) and a control group (CG; n=14).

The experimental group will perform the 'Odd One Out', 'Double Trouble', and 'Monkey Ladder' tests immediately before and after a hypoxia tolerance session (12% oxygen, equivalent to 4400 meters) using the iAltitude simulator. The control group will complete the same tests under normoxic conditions, without exposure to hypoxia.

The primary outcomes will include changes in cognitive performance scores in the administered tests. The experimental group is expected to show improvements in the Double Trouble test scores following hypoxia exposure. The control group may also show changes in the Double Trouble and Odd One Out tests between the pre- and post-tests.

Secondary outcomes will include physiological variables such as oxygen saturation (SaO₂) and heart rate (HR), which will be monitored during the hypoxia session in the EG. Statistically significant changes in SaO₂ and HR are anticipated as a result of the hypoxic exposure.

This study aims to determine whether a single session of intermittent normobaric hypoxia can lead to selective improvements in executive functions, particularly sustained attention, without negatively affecting other cognitive domains.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged between 18 and 40 years old

Exclusion Criteria:

* Pregnancy
* Prior experience in hypoxia training
* Previous experience in executive function tests
* Personal or family history of cardiovascular diseases or chronic conditions
* Diagnosed cardiac disorders.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Double Trouble Test | Day 1
  Change in cognitive performance score on the Double Trouble test; higher scores indicate better executive function and attention control. Unit of Measure: Score (units on a scale)
Monkey Ladder Test | Day 1
  Change in cognitive performance score on the Monkey Ladder test; higher scores indicate better visuospatial working memory. Unit of Measure: Score and Level.
Odd One Out Test | Day 1
  Change in reasoning performance score on the Odd One Out test; higher scores indicate better problem-solving ability. Unit of Measure: Score and Level.

SECONDARY OUTCOMES:
Blood Pressure | Day 1
  Average of systolic and diastolic blood pressure measured in mmHg
Oxygen Saturation | During intervention
  Oxygen saturation automatically monitored and recorded by the iAltitude hypoxia simulation system. Unit of Measure: %
Heart Rate | During intervention
  Heart rate automatically monitored and recorded by the iAltitude hypoxia simulation system. Unit of Measure: Beats per minute (bpm)
Sociodemographic Questionnaire | Pre-test
  To define individual characteristics of participants such as age and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Raquel Vaquero Cristóbal, PhD, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (2):
- Spain (2):
  - Universidad Católica San Antonio de Murcia, Murcia, Guadalupe
  - Universidad Católica San Antonio de Murcia, Murcia

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to ethical and privacy considerations.